CLINICAL TRIAL: NCT05422703
Title: Combined Effect of Manual Therapy and Kinesio Taping on Temporomandibular Joint Dysfunction Following Oral Surgeries
Brief Title: Manual Therapy and Kinesio Taping on Temporomandibular Joint Dysfunction Following Oral Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Kamal Mousa Mohamed, Combined effect of manual therapy and kinesiotaping on temporomandibular joint dysfunction following oral surgeries, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/003508
Record Dates: First submitted 2022-06-10; First posted 2022-06-16 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Temporomandibular Joint Dysfunction
Keywords: Kinesio taping; Manual therapy; Oral surgeries
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Athletic Tape; Musculoskeletal Manipulations; Exercise; Analgesics; Peptide Hydrolases; Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): patients who will receive manual therapy and Kinesio taping, in additional to basic post operative care (ice pack , analgesics, Antibiotic treatment and mouth wash daily ) 3 times per week for two weeks.
  Interventions: Device: Kinesio tape; Other: Gauze pack; Device: ice pack; Procedure: Manual therapy; Drug: Analgesic; Drug: Proteolytic enzymes; Drug: Mouth wash; Dietary Supplement: Soft cold diet
- Control group (Placebo Comparator): patients who will receive basic post operative care (ice pack , analgesics, Antibiotic treatment and mouth wash daily ).
  Interventions: Other: Gauze pack; Device: ice pack; Drug: Analgesic; Drug: Proteolytic enzymes; Drug: Mouth wash; Dietary Supplement: Soft cold diet

INTERVENTIONS:
Device: Kinesio tape — Skin-colored Kinesiology Tape (ARES tape,5 cm×5 m) is waterproof tape is made of 100% cotton,applied in the shape of a fan strip, waterproof. The width is 5 cm and thickness of 0.5 mm (5 cm×5 m ).This tape is sticking with a small stretch (about 15%).
  Arms: Study group
Other: Gauze pack — Place gauze pack over surgical site for one hour after surgery.
Device: ice pack — Ice packs will be applied for 6 hours after surgery in all patients
Procedure: Manual therapy — passive and active range of motion, stretching exercises, resistive mouth exercises, mobilization exercises and coordination exercices.
  Other Names: Exercises
  Arms: Study group
Drug: Analgesic — NSAIDs like ibuprofen (600-800 mg) or declophenac sodium (50-150 mg) 3 times a day
Drug: Proteolytic enzymes — 1-2 ampoules daily IM box of 3 ampoules of 5 mg crystallized and lyophilized chymotrypsin (450 E. A. Units) + 3 ampoules of 3 ml apyrogenic saline for one week.
Drug: Mouth wash — use 0.12% chlorhexidine or povidone iodine mouthwash daily
Dietary Supplement: Soft cold diet — For the day of surgery

SUMMARY:
Oral surgeries include various types such as impacted wisdom tooth surgery, oral cyst enucleation (cystectomy), surgical incision and drainage of odontogenic abcess, oral tumor excision and open reduction and internal fixation of mandibular fracture (ORIF). Oral surgeries are usually associated with pain, swelling and inability to open the mouth. Those symptoms reach the maximum intensity between the third to fifth days postoperatively for the swelling and 24 to 48 hours postoperatively for the pain and then, they gradually diminished until the 7th day postoperatively

DETAILED DESCRIPTION:
Oral surgery concerned with the diagnosis and surgical treatment of congenital or acquired diseases, dysfunction, defects or injuries of the mouth and jaw. Oral surgeries include various types such as impacted wisdom tooth surgery, oral cyst enucleation (cystectomy), surgical incision and drainage of odontogenic abscess, oral tumor excision and open reduction and internal fixation of mandibular fracture (ORIF).

Temporomandibular joint dysfunction: It is one of post operative complications that occur post oral surgeries which include several symptoms as pain,edema and trismus. Pain is the most common and limiting clinical manifestation of this dysfunction, as well as decreased mobility of the jaw, both of which impacts quality of life. The multifactor etiology of temporomandibular joint dysfunction often requires multidisciplinary healthcare professionals to manage difficult symptoms, including chronic pain. Many studies have identified a variety of conservative interventions, such as physical therapy, for patients with temporomandibular joint disorders, including joint mobilization, tissue mobilization,dry needling, friction massage, patient education, splints, modalities, stretching, coordination activities,strengthening exercises, and combinations of these techniques. postoperative major complications such as pain, edema and trismus in various oral surgeries such as tooth extraction, maxillary expansion, and orthognathic surgeries. Oral surgical procedures are often accompanied by a multitude of complications including pain, swelling, and morbidity. These are the result of inflammatory processes induced by the surgical wound healing.

Facial edema: During surgeries, inflammatory chemicals such as prostaglandins, leukotrienes, bradykinins, and platelet-activation factors are secreted by damaged tissue. Moreover, excessive lymph production causes disturbances in local lymphatic circulation. Inflammatory chemicals create endothelial gaps to increase vascular permeability. In addition, macrophages and mast cells in damaged tissues produce histamine, serotonin, and eicosanoids; alter the local constitution of blood vessels; and release nitric oxide, eventually resulting in vasorelaxation. These chain reactions increase blood vessel relaxation and vascular permeability and result in the accumulation of interstitial fluid, eventually resulting in tissue swelling and pain.

Trismus: It is defined as prolonged tetanic spasm of masticatory muscles of jaw. the transient jaw stiffness usually reaches its peak on the 2nd day post surgery. It is diagnosed from clinical examination of the maximal interincisal distance (MID) <40-45 mm caused by contracture and not by obstructive joint impingement.The factors contributing to trismus are: (1) Multiple needle penetrations correlate with a greater incidence of post injection trismus. (2) Elevation of flap beyond the external oblique ridge. (3) At times, the patient hurts his/her own tongue or cheek under the effect of anesthesia resulting in reflex trismus.

kinesio taping (KT) was developed by the Japanese therapist and academic lecturer. More than 30 years ago, he created a special tape, which by the correct application, i.e. sticking with a small stretch (about 15%) to the skin, raises the surface of the skin, thereby increasing the space between the dermis and fascia . The expansion of this space, should reduce lymph retention. The patch used for this method has a thickness and weight similar to skin. The waterproof tape is made of 100% cotton, while the adhesive on the inside is applied in the shape of a fan strip, which allows the air to flow. When stretched beyond its normal length and applied, it recoils and creates a pulling force on the skin, thus improving blood and lymph flow by alleviating hemorrhage and congestion of lymphatic fluid.

Manual therapy (MT) is one of the various types of interventions for treating patients with temporomandibular joint dysfunction and include: Mobilization exercise stretching exercise, coordination exercise, rang of motion exercise and strengthening exercise. Within other body regions, manual therapy intervention has been detailed and summarize the efficacy of treatment approaches.Strengthening, stretching/flexibility, and motor control exercises have demonstrated to be efficacious in reducing pain and disability in patients with chronic low back pain,as well as mechanical neck pain. Despite a review and meta-analysis the efficacy of exercise therapy and dosage has yet to be determined for patients with temporomandibular joint dysfunction. exercises intended to increase mobility of the temporomandibular joint and/or muscles of the jaw. Exercise therapy aims to reduce clinical symptoms such as pain in the muscles and joints, and improve motor function by moving whole or part of the body.Exercise can be classified into self exercise by patients and manual therapy that physiotherapists apply to patients. Self exercise is often offered as home exercise or self-care program that can be done at home. manual exercise therapy includes mobilization, stretch,muscle strengthening exercise and coordination exercise.

ELIGIBILITY:
Inclusion Criteria:

* age ranged between 20-50 years
* both gender
* TMJ dysfunction following oral surgeries.

Exclusion Criteria:

* open wound in affected area
* facial trauma,smoker and infection
* sensitivity to tape
* allergies to medication administered in the study
* reluctance to shave facial hair (for men)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
facial swelling | Two weeks
  Facial swelling was assessed by a four-line measurement method using a flexible plastic tape measure. The corresponding lines were line A from the most posterior point of the tragus to the most lateral point of the lip commissure),line B (from the most posterior point of the tragus to the pogonion), line C from the most inferior point of the mandibular angle to lateral canthus of the eye ; and line D, most inferior point of the mandibular angle to (the nasal border - wing of the nostril. These measurements were performed with the patient sitting at 90° straight position with physiologic rest position of the mandible.
Facial pain | Two weeks
  Visual analogue scale (VAS)measure, consists of a line usually 10 cm in length, with anchor descriptors such as (in the pain context) where 0 means no pain and 10 means worst conceivable pain. patients asked to mark the point corresponding to the intensity of their pain , and the distance from the left endpoint to the mark is measured, in cm.
Maximum mouth opening | Two weeks
  measurement of maximal interincisal distance (mm) attained during the active mouth opening by the subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lietz-Kijak D, Kijak E, Krajczy M, Bogacz K, Luniewski J, Szczegielniak J. The Impact of the Use of Kinesio Taping Method on the Reduction of Swelling in Patients After Orthognathic Surgery: A Pilot Study. Med Sci Monit. 2018 Jun 4;24:3736-3743. doi: 10.12659/MSM.909915. PMID 29861496
- [Background] Yurttutan ME, Sancak KT. The effect of kinesio taping with the web strip technique on pain, edema, and trismus after impacted mandibular third molar surgery. Niger J Clin Pract. 2020 Sep;23(9):1260-1265. doi: 10.4103/njcp.njcp_23_20. PMID 32913166
- [Background] Jaron A, Preuss O, Grzywacz E, Trybek G. The Impact of Using Kinesio Tape on Non-Infectious Complications after Impacted Mandibular Third Molar Surgery. Int J Environ Res Public Health. 2021 Jan 6;18(2):399. doi: 10.3390/ijerph18020399. PMID 33419167
- [Background] Tatli U, Benlidayi IC, Salimov F, Guzel R. Effectiveness of kinesio taping on postoperative morbidity after impacted mandibular third molar surgery: a prospective, randomized, placebo-controlled clinical study. J Appl Oral Sci. 2020;28:e20200159. doi: 10.1590/1678-7757-2020-0159. Epub 2020 Jul 13. PMID 32667383